CLINICAL TRIAL: NCT01867671
Title: Oral Immunotherapy for Induction of Tolerance and Desensitization in Peanut-Allergic Children (ITN050AD)
Brief Title: Peanut Oral Immunotherapy in Children
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ITN050AD
Record Dates: First submitted 2013-05-23; First posted 2013-06-04 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Peanut Hypersensitivity
Keywords: Allergy, Peanut; Peanut allergy; Hypersensitivity; Immunotherapy; Desensitization, Immunologic
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut Oral Immune Therapy (OIT) (Experimental): Peanut OIT for 134 weeks followed by peanut avoidance for 26 weeks.
  Interventions: Biological: Peanut Oral Immunotherapy - Liquid Extract; Biological: Peanut Oral Immunotherapy - Peanut Flour
- Peanut Placebo (Placebo Comparator): Peanut placebo for 134 weeks followed by peanut avoidance for 26 weeks. The placebo extract will be derived from oat flour source material.
  Interventions: Biological: Placebo for Peanut Oral Immunotherapy - Liquid Extract form; Biological: Placebo for Peanut Oral Immunotherapy - Peanut Flour

INTERVENTIONS:
Biological: Peanut Oral Immunotherapy - Liquid Extract — Used during initial dose escalation for doses 0.1 to 0.8 mg.
  Arms: Peanut Oral Immune Therapy (OIT)
Biological: Placebo for Peanut Oral Immunotherapy - Liquid Extract form — Similar in appearance, texture, and taste to peanut liquid extract.
  Arms: Peanut Placebo
Biological: Peanut Oral Immunotherapy - Peanut Flour — This will be used for the remainder of dose escalation, build-up, and maintenance.
  Arms: Peanut Oral Immune Therapy (OIT)
Biological: Placebo for Peanut Oral Immunotherapy - Peanut Flour — Similar in appearance, texture, and taste to peanut flour.
  Arms: Peanut Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center study comparing peanut oral immunotherapy (OIT) to placebo in the induction of tolerance and desensitization in peanut-allergic children. Eligible participants with peanut allergy will be randomly assigned to receive either peanut OIT or placebo for 134 weeks followed by peanut avoidance for 26 weeks.

DETAILED DESCRIPTION:
An initial oral food challenge (OFC) to 1 g of peanut flour (500 mg peanut protein) will be conducted. Participants must have a clinical reaction during this OFC to initiate study dosing. After the initial OFC, the study design includes four phases:

* Initial dose escalation (1 day): Peanut or placebo dosing will be given incrementally and increase every 20 minutes until a dose of 12 mg peanut flour (6 mg peanut protein) or placebo flour is given.
* Build-up (30 weeks): Initial observed dose administration of highest tolerated dose, followed by daily OIT at home with return visit every 2 weeks for dose escalation.
* Maintenance (104 weeks):The participant will continue on daily OIT with return visits every 13 weeks. At the end of this phase the participant will undergo a blinded OFC to 10 g peanut flour (5 g peanut protein).
* Avoidance (26 weeks): In this final phase participants will be seen every 13 weeks. At the completion of this phase participants will have a final blinded OFC to 10g peanut flour (5 g peanut protein).

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of peanut allergy or avoidance of peanut without ever having eaten peanut;
* Serum immunoglobulin E (IgE) to peanut of ≥5 kUA/L determined by UniCAP™, an in-vitro test system for diagnosis and monitoring of allergy and inflammation;
* Wheal ≥ 3mm on skin prick test to peanut extract compared to a negative control;
* A clinical reaction at or below ingestion of 1 g peanut flour (500 mg peanut protein) during screening OFC;
* Written informed consent from parent/guardian.

Exclusion Criteria:

* History of severe anaphylaxis with hypotension to peanut;
* Documented clinical history of allergy to oat;
* Suspected allergy to oat and a wheal ≥7mm on skin prick test to oat extract compared to a negative control;
* Chronic disease other than asthma, atopic dermatitis, rhinitis requiring therapy; e.g., heart disease or diabetes;
* Active eosinophilic gastrointestinal disease in the past 2 years;
* Participation in any interventional study for the treatment of food allergy in the 6 months prior to visit -1;
* Inhalant allergen immunotherapy that has not yet reached maintenance dosing;
* Severe asthma, as indicated by repeated hospitalizations or hospital emergency department visits;
* Moderate asthma defined according to National Asthma Education and Prevention Program Expert;
* Panel that requires more than fluticasone 440 mcg or its equivalent daily for adequate control;
* Inability to discontinue antihistamines for skin testing, OFC and the initial dose escalation;
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) in the 12 months prior to visit -1;
* Any systemic therapy which in the judgment of the investigator could be immunomodulatory (e.g. rituximab) in the 12 months prior to visit -1, systemic corticosteroid therapy of up to a total of three weeks is allowed;
* Use of any investigational drug in 90 days prior to visit -1;
* Plan to use any investigational drug during the study period;
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Study Chair — UNC Chapel-Hill; Stacie M. Jones, MD, Study Chair — University of Arkansas
Locations (5):
- United States (5):
  - University of Arkansas for Medical Sciences: Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University School of Medicine, Stanford, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York
  - UNC Chapel-Hill, Chapel Hill, North Carolina

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: ITN IMPACT Study website — http://www.impactstudy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ages 1 to 3 with a clinical history of peanut allergy or avoidance of peanut without ever having eaten peanut were recruited from 5 clinical centers in the United States from August 2013 to October 2015.
Pre-assignment Details: Individuals with a history of severe anaphylaxis (previous hypotension) to peanut were excluded.
Groups:
- Peanut Oral Immune Therapy (OIT): Peanut Oral Immune Therapy (OIT) for 134 weeks followed by peanut avoidance for 26 weeks.
  Two forms of peanut oral immunotherapy were used. One form was a liquid extract derived from the peanut flour source material. This was used during initial dose escalation for doses 0.1 to 0.8 mg of peanut protein. The second form was peanut flour, which was used for the remainder of dose escalation, build-up, and maintenance.
- Peanut Placebo: Peanut placebo for 134 weeks followed by peanut avoidance for 26 weeks.
  Two forms of placebo were used. One form was a liquid extract derived from oat flour source material. This was used during initial dose escalation for doses 0.1 to 0.8 mg. The second form was peanut flour, which was used for the remainder of dose escalation, build-up, and maintenance.
Period: Overall Study
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo
Started | 96 | 50
Completed | 67 | 22
Not Completed | 29 | 28
Not completed — Adverse Event | 5 | 3
Not completed — Anaphylaxis | 0 | 1
Not completed — Inability to reach 3 mg peanut/placebo | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with Study Drug | 1 | 2
Not completed — Withdrawal by Subject | 21 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo | Total
Number analyzed (Participants) | 96 | 50 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (0.7) | 3.0 (0.8) | 3.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 18 | 48
  Male | 66 | 32 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 92 | 45 | 137
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 64 | 31 | 95
  More than one race | 16 | 11 | 27
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 96 | 50 | 146

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Desensitized to Peanut Protein After 134 Weeks of Oral Immunotherapy (OIT)
Description: Definition of desensitized to peanut: A participant who passed the blinded (masked) oral food challenge (OFC) to10 grams of peanut flour (=5 grams of peanut protein) without significant symptoms.*
  *Significant symptoms include hives, wheezing, vomiting, or laryngeal edema.
Time Frame: Week 134
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo
Number analyzed (Participants) | 96 | 50
Percentage of Participants | 71 [61.7 to 79.9] | 2 [0.0 to 5.9]
Statistical Analysis 1: Comparison: Peanut Oral Immune Therapy (OIT) vs Peanut Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 205.45, 95% CI 2-sided [24.00 to 1758.51]

2. Secondary Outcome: Percentage of Tolerant Participants at Week 160
Description: Definition of Tolerant: A participant who passed the oral food challenge (OFC) to 10 grams of peanut flour (=5 grams of peanut protein).
Time Frame: Week 160
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo
Number analyzed (Participants) | 96 | 50
percentage of participants | 21 [12.7 to 29.0] | 2 [0.0 to 5.9]
Statistical Analysis 1: Comparison: Peanut Oral Immune Therapy (OIT) vs Peanut Placebo; Test type: Superiority; p < 0.0031, Regression, Logistic; Odds Ratio (OR) = 27.82, 95% CI 2-sided [3.07 to 252.33]

3. Secondary Outcome: Count of Participants With Transient Desensitization
Description: Definition of transient desensitization: A participant who passed the blinded (masked) oral food challenge (OFC) to 10 grams peanut flour (=5 grams peanut protein) at week 134 and failed the week 160 in the Peanut oral immunotherapy (OIT) group.
Time Frame: Week 134, Week 160
Population: Participants randomized to the Peanut Oral Immunotherapy (OIT) group
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Oral Immune Therapy (OIT)
Number analyzed (Participants) | 96
Participants
  Passed Week 134 and Failed Week 160 | 49
  Passed Week 134 and Passed Week 160 | 19
  Failed Week 134 and Failed Week 160 | 27
  Failed Week 134 and Passed Week 160 | 1
Statistical Analysis 1: Comparison: Peanut Oral Immune Therapy (OIT); Test type: Other — McNemar's Test; p < 0.0001, McNemar; Simple Kappa Coefficient = 0.1620, 95% CI 2-sided [0.0628 to 0.2612]

4. Secondary Outcome: Highest Tolerated Cumulative Dose
Description: The highest tolerated cumulative dose of peanut protein during the blinded (masked) oral food challenge (OFC) at Week 160, analyzed within and between both placebo and peanut OIT groups. The highest cumulative dose of peanut protein tolerated for each participant was analyzed as a continuous outcome.
  Any randomized participant without an evaluable blinded (masked) OFC was imputed as not tolerant. For the continuous highest cumulative dose endpoint, this is defined as having a highest cumulative dose imputed as zero.
Time Frame: Week 160
Measure: Mean (95% Confidence Interval); unit: mg protein
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo
Number analyzed (Participants) | 96 | 50
mg protein | 1645 [1338 to 1951] | 180 [-244 to 605]
Statistical Analysis 1: Comparison: Peanut Oral Immune Therapy (OIT) vs Peanut Placebo; Test type: Superiority; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 1464, 95% CI 2-sided [944 to 1985]

5. Secondary Outcome: Percentage of Participants That Withdrew From the Study
Description: Percentage of participants that withdrew from study participation, listed by study phase (at time of study withdrawal).
Time Frame: Initial Dose Escalation through Week 160 (Tolerance Assessment)
Measure: Number; unit: percentage of participants
Arm/Group | Peanut Oral Immune Therapy (OIT) | Peanut Placebo
Number analyzed (Participants) | 96 | 50
percentage of participants
  Terminated during Initial Dose Escalation | 2 | 0
  Terminated during Build-Up | 4 | 12
  Terminated during Maintenance | 8 | 16
  Terminated after Maintenance/Prior to OFC | 1 | 2
  Terminated during Avoidance | 11 | 14
  Terminated after Avoidance/Prior to OFC | 0 | 10
  Terminated after Tolerance Assessment | 3 | 2

ADVERSE EVENTS:
Time Frame: 162 weeks
Groups:
- Peanut Oral Immunotherapy (OIT): Peanut OIT for 134 weeks followed by peanut avoidance for 26 weeks.
- Peanut Placebo: Peanut placebo for 134 weeks followed by peanut avoidance for 26 weeks. The placebo extract was derived from oat flour source material.
Arm/Group | Peanut Oral Immunotherapy (OIT) | Peanut Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/96 | 4/50
Other Adverse Events (participants affected / at risk) | 96/96 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut Oral Immunotherapy (OIT) (N=96) | Peanut Placebo (N=50)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut Oral Immunotherapy (OIT) (N=96) | Peanut Placebo (N=50)
Ear pain (Ear and labyrinth disorders) | 4 (9) | 3 (3)
Conjunctivitis (Eye disorders) | 6 (8) | 5 (9)
Abdominal discomfort (Gastrointestinal disorders) | 18 (48) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 29 (105) | 5 (18)
Abdominal pain upper (Gastrointestinal disorders) | 10 (26) | 2 (4)
Constipation (Gastrointestinal disorders) | 8 (8) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 20 (26) | 12 (20)
Gastritis (Gastrointestinal disorders) | 13 (19) | 5 (15)
Lip pruritus (Gastrointestinal disorders) | 5 (10) | 0 (0)
Vomiting (Gastrointestinal disorders) | 45 (80) | 19 (32)
Influenza like illness (General disorders) | 20 (78) | 8 (27)
Pyrexia (General disorders) | 65 (190) | 29 (108)
Allergy to animal (Immune system disorders) | 6 (15) | 3 (6)
Food allergy (Immune system disorders) | 85 (135) | 43 (72)
Hypersensitivity (Immune system disorders) | 39 (77) | 15 (25)
Type I hypersensitivity (Immune system disorders) | 75 (1047) | 31 (152)
Bronchitis (Infections and infestations) | 3 (3) | 3 (4)
Croup infectious (Infections and infestations) | 14 (27) | 5 (7)
Ear infection (Infections and infestations) | 12 (14) | 7 (8)
Gastroenteritis (Infections and infestations) | 35 (48) | 12 (19)
Gastroenteritis viral (Infections and infestations) | 19 (27) | 9 (9)
Hand-foot-and-mouth disease (Infections and infestations) | 6 (6) | 2 (2)
Impetigo (Infections and infestations) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 8 (9) | 7 (7)
Molluscum contagiosum (Infections and infestations) | 5 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (13) | 2 (8)
Otitis media (Infections and infestations) | 23 (38) | 15 (21)
Otitis media acute (Infections and infestations) | 5 (5) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 21 (28) | 3 (8)
Pneumonia (Infections and infestations) | 9 (10) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Sinusitis (Infections and infestations) | 13 (19) | 5 (16)
Upper respiratory tract infection (Infections and infestations) | 34 (73) | 18 (42)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Viral infection (Infections and infestations) | 33 (67) | 12 (16)
Viral upper respiratory tract infection (Infections and infestations) | 26 (42) | 8 (14)
Excoriation (Injury, poisoning and procedural complications) | 1 (2) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Headache (Nervous system disorders) | 8 (11) | 1 (1)
Agitation (Psychiatric disorders) | 9 (10) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (133) | 23 (49)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 (39) | 9 (18)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 20 (33) | 6 (17)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 17 (33) | 15 (22)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 9 (13) | 7 (8)
Eczema (Skin and subcutaneous tissue disorders) | 27 (65) | 12 (16)
Erythema (Skin and subcutaneous tissue disorders) | 5 (8) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (39) | 10 (17)
Rash (Skin and subcutaneous tissue disorders) | 24 (33) | 11 (24)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 24 (65) | 16 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT01867671/Prot_SAP_000.pdf